CLINICAL TRIAL: NCT05656131
Title: Fluzoparib in Combination With or Without Camrelizumab for Homologous Recombinant Deficiency (HRD) HER2 Negative Advanced Breast Cancer，A Two-cohort, Open, Multicenter，Phase II Study
Brief Title: Fluzoparib in Combination With or Without Camrelizumab for Homologous Recombinant Deficiency (HRD) HER2 Negative Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: wang shusen (Other)
Responsible Party: Sponsor-Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-042
Record Dates: First submitted 2022-12-11; First posted 2022-12-19 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Advanced HER2 Negative Breast Carcinoma HRD+Breast Cancer
MeSH Terms: interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluzoparib (Experimental): Fluzoparib: 150 mg twice daily (morning and evening) for 21 consecutive days as a cycle until disease progression or intolerance.
  Interventions: Drug: Fluzoparib
- fluzoparib+Camrelizumab (Experimental): Fluzoparib: 150 mg twice daily (morning and evening) for 21 consecutive days as a cycle until disease progression or intolerance.
  Camrelizumab: 200 mg IV drip over approximately 30 minutes (no less than 20 minutes and no more than 60 minutes) on Day 1 of each 3-week treatment cycle until disease progression or intolerance.
  Interventions: Drug: Fluzoparib+Camrelizumab

INTERVENTIONS:
Drug: Fluzoparib — Arms A will be treated with fluzoparib alone
  Arms: fluzoparib
Drug: Fluzoparib+Camrelizumab — Arms B will be treated with fluzoparib in combination with camrelizumab
  Arms: fluzoparib+Camrelizumab

SUMMARY:
This study is planned to include 80 patients with HRD positive HER2-negative advanced breast cancer to receive fluzoparib alone or fluzoparib combined with camrelizumab to observe and evaluate the efficacy and safety of fluzoparib combined with or without camrelizumab in the treatment of HRD positive HER2-negative advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years old
2. Histologically or cytologically confirmed locally advanced or metastatic breast cancer.
3. Pathologically documented breast cancer that is HER2-negative for both primary tumor and metastases (if puncture results are available)
4. ECOG PS of 0-1.
5. For locally advanced or metastatic breast cancer, the tumor tissue HRD score> 42 is needed (for HRD testing, the recipient must provide a test report from an institution with a qualified testing unit prior to enrollment; if no report is available, the relevant test sample must be provided for confirmation in the central laboratory prior to enrollment).
6. Presence of at least 1 measurable lesion based on computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1).
7. If treated with PARP inhibitors or immune checkpoint inhibitors in the (neo) adjuvant phase, a relapse-free interval of more than 1 year after the end of treatment is required.
8. Prior treatment with paclitaxel-based chemotherapeutic agents is allowed.
9. ≤ 2 lines of prior chemotherapy in the advanced stage.
10. For HR+ patients, progression within two years of (neo) adjuvant endocrine therapy is required; patients who have progressed after more than two years of endocrine therapy are required to have received at least first-line endocrine therapy for metastatic disease (including CDK4/6 inhibitors, cidarabine and PI3K inhibitors, etc.).
11. ≤ grade 1 (CTCAE v5.0) for all toxicities occurring in relation to prior antitumor therapy. However, patients with any grade of alopecia are allowed to enter the study.
12. CNS metastases without symptoms may be enrolled.

    * If there is no extracranial assessable lesion, intracranial lesions are required to be assessable and suitable for systemic therapy only
    * If there is an extracranial evaluable lesion, patients with an intracranial lesion that has been stabilized with local therapy may be accepted for enrollment
13. Routine blood tests within 1 week prior to enrollment are essentially normal.

    * White blood cell count (WBC) ≥ 2.5 × 109/L.
    * Neutrophil count (ANC) ≥ 1.5 × 109/L.
    * Platelet count (PLT) ≥ 75 × 109/L.
    * Patients may receive blood transfusions or erythropoietin therapy to meet this criterion.
14. Basic normal liver and renal function tests within 1 week prior to enrollment.

    * Total bilirubin (T BIL) ≤ 1.5 x the upper limit of normal (ULN).
    * Glutathione transaminase (SGPT/ALT) ≤ 2.5 x ULN (≤ 5 x ULN in patients with liver metastases).
    * Glutathione aminotransferase (SGOT/AST) ≤ 2.5× ULN (≤ 5× ULN in patients with liver metastases).
    * creatinine clearance (Ccr) ≥ 60 ml/min.
15. Patients subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and after the last dose of treatment medicine for at least 90 days.
16. A life expectancy of at least 12 weeks.
17. Patients must be able to participate and comply with treatment and follow-up.

Exclusion Criteria:

1. Has multiple primary malignancies and requires standardized treatment or major surgery within 2 years of the first dose of study treatment.
2. Treated with PARP inhibitors in advanced stages.
3. BRCA1/2 germline mutation.
4. Symptomatic or unstable brain metastases.
5. Any severe or poorly controlled systemic disease such as poorly controlled hypertension, active bleeding susceptibility or active infection, as judged by the investigator. Chronic disease needs to be excluded.
6. Refractory nausea, vomiting or chronic gastrointestinal disease, inability to swallow study drug or previous extensive bowel resection that may interfere with adequate absorption of PARP inhibitors.
7. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, interstitial lung disease, pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion etc), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjögren's, sarcoidosis etc), or prior pneumonectomy.
8. Otherwise considered inappropriate for the study by the Investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 3 years
  Objective response is defined as a complete response (CR) or partial response (PR) according to RECIST v.1.1.recorded from randomization until disease progression or death due to any cause

SECONDARY OUTCOMES:
Progress-free survival | Up to 3 years
  Time from randomization to the first documentation of objective tumor progression or to death due to any cause
Overall Survival | Up to 3 years
  Time from randomization to date of death due to any cause. according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death to any cause.
QoL questionnaire （quality of life） | Up to 3 years
Adverse effect (AE) | Up to 3 years
  Any adverse effect occurred in the treatment

CONTACTS AND LOCATIONS:
Overall Officials: shusen Wang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun-yat sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No